CLINICAL TRIAL: NCT04850482
Title: Feasibility Randomised Controlled Trial of the MyJourney Web App, Supporting Adjustment to an Unfulfilled Wish for Children.
Brief Title: Feasibility Trial of the MyJourney Web App: Supporting Adjustment to an Unfulfilled Wish for Children.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Cardiff University (Other)
Collaborators: Portuguese Fertility Association (Unknown); Fertility Network UK (Unknown)
Responsible Party: Principal Investigator, Sofia Gameiro, Principal Investigator, Cardiff University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: EC.20.10.13.6082
Record Dates: First submitted 2021-01-13; First posted 2021-04-20 (Actual); Last update posted 2021-08-03 (Actual); Status verified 2021-08

CONDITIONS: Mental Health
Keywords: Well being; Unfulfilled wish for children; Self-Help; Online intervention; Involuntary childlessness
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: Two arm, parallel-group, non-blind feasibility trial with 1:1 allocation to the intervention group (immediate access to MyJourney) or waitlist control group (receives access to MyJourney after 10 weeks).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Arm (Experimental): Participants get immediate access to the intervention on completion of baseline assessment.
  Interventions: Other: MyJourney
- Wait list control Arm (No Intervention): Participants get access to the intervention in 10 weeks after completion of the baseline and follow up assessment.

INTERVENTIONS:
Other: MyJourney — MyJourney is an online self-help interactive program based on Contextual Cognitive Behavioural Therapy.
  Arms: Intervention Arm

SUMMARY:
A bilingual online self-help app - MyJourney - has been developed for individuals faced with an unfulfilled wish for children. The specific aim of this trial is to evaluate the feasibility, defined here as determining whether the intervention itself and the study procedures are appropriate for further evaluation, and how users react to the intervention, which will inform the implementation of a future full scale RCT to evaluate MyJourney's efficacy.

This RCT will be a two arm, parallel-group, non-blind feasibility trial with 1:1 allocation to the intervention group (immediate access to MyJourney) or waitlist control group (receives access to MyJourney after 10 weeks). A minimum number of 152 individuals will be enrolled in this study. Once participants have met the eligibility criteria and completed the baseline assessment, they will be randomly assigned to one of two groups: the intervention group or the waitlist control group. The sample will be recruited online.

Participation in this study will last 10 weeks for the waitlist group and 6 months for the intervention group. Participants in both groups will be invited to complete a baseline assessment (online survey) and a follow-up assessment (online survey) at 10-weeks post baseline. The intervention group will also be invited to complete another follow-up assessment at 6-months post baseline. Assessments will include self-report questionnaires to cover socio-demographic information (baseline only), psychological mediators (mechanisms of change) (baseline and 10-week follow-up), psychological outcome questionnaires (baseline, 10-week and 6-month follow up), and questions about acceptability and feasibility (10-week and 6-month follow up).

DETAILED DESCRIPTION:
In this trial, a bilingual self-help web-app, MyJourney, developed to support individuals with an unfulfilled wish for children, will be evaluated for feasibility. This trial forms part of the exploratory trial phase of development of complex interventions, based on guidance from the Medical Research Council.

Although research has demonstrated that those faced with an unfulfilled wish for children (i.e., the inability to have all the children desired) can experience intense grief and worse mental health for a prolonged period, at present there is limited evidence for a theory led intervention that would provide support for this group and to date there is no widely used evidence-based interventions for individuals facing an unfulfilled wish for children. An in-depth systematic review of how people adjust to an unfulfilled wish for children informed the Three Task Model (3TM). This proposes three psychological mechanisms that facilitate adjustment to an unfulfilled wish for children: acceptance, meaning making and pursuit of new life goals, leading to better mental-health and well-being.

Therefore, a bilingual online self-help web app - MyJourney - was developed. The 3TM informed the hypothesised mechanisms of the change targeted by the intervention. Contextual Cognitive Behavioural Therapy (CCBT) was chosen as the therapeutic framework for each of the steps within the intervention, focussing on a person's relationships with their thoughts, emotions and behaviours. The intervention consists of 10 ordered Steps. Each Step is a structured therapeutic activity designed to activate a specific technique which is linked to the theorized mechanism of change. Each Step has up to three optional therapeutic resources designed to encourage participants to engage with and practice the therapeutic skill they are developing. Users are invited to engage with one Step per week over 10 weeks, however they are able to engage at their own pace.

The specific aim of this trial is to evaluate feasibility, defined here as determining whether the intervention itself and the study procedures are appropriate for further evaluation, and how users react to the intervention, which will inform the implementation of a future full scale RCT to evaluate MyJourney's efficacy. Several feasibility outcomes will be focussed on, including acceptability, demand, implementation, practicality, adaption, and limited efficacy testing. In addition, the targeted mechanisms of change will also be evaluated.

This RCT will be a two arm, parallel-group, non-blind feasibility trial with 1:1 allocation to the intervention group (immediate access to MyJourney) or waitlist control group (receives access to MyJourney after 10 weeks). There will be three assessment moments: one at baseline (pre-exposure to intervention); 10 weeks after baseline (post exposure to intervention); and 6 months after baseline (intervention group only).

Participants will be recruited via appropriate websites, social media, blogs, via direct contact with appropriate support groups and Prolific. A minimum of 50 participants will be required, and accounting for participation and attrition rates, a minimum of 152 individuals need to be recruited.

Participants will be directed to https://myjourney.pt from the trial advertisements and upon clicking 'Get Started' will be informed of the trial goals, structure and participant roles. Individuals who decided to take part in the trial will be provided with an information sheet and they will then give their informed consent. One they have indicated their eligibility and completed the baseline assessment (socio-demographic details, psychological mediators and outcomes), they will be randomly assigned to the intervention group or the waitlist control group. The participants assigned to the waitlist control will be informed that they are on a waiting-list and that they will receive access to the MyJourney in 10 weeks. The participants in the intervention group will be provided with a link to register to MyJourney.

Ten weeks after completion of the baseline assessment, participants in the intervention and waitlist control groups will be invited to complete a follow up assessment. The ten-week follow-up assessment will ask participants to report on psychological mediators and outcomes and the intervention group will complete a section on acceptability of MyJourney. At the end of completing this assessment, participants in the waitlist control group will be provided with a debrief form and given access to MyJourney. Six months after baseline, participants in the intervention group (only) will be invited to complete another follow up assessment covering only psychological outcomes, at the end of which they will be provided with a debrief form. Some participants will also take part in an interview as part of the study's process evaluation.

ELIGIBILITY:
Inclusion Criteria:

* able to provide consent
* self-identifying as having an unfulfilled wish for children
* being able to use and access MyJourney (have an internet connection, suitable device and have an active email address)
* speak English or Portuguese
* be able to fill out online questionnaires

Exclusion Criteria:

* diagnosed with a mental-health disorder within the last 2 years [self-reported]
* currently receiving therapy for a clinically diagnosed mental-health disorder
* individual or group therapy or peer support specifically related to their unfulfilled wish for children [self-reported]
* unable to use MyJourney due to other health problems (e.g., vision impairments)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 221 (Actual)
Dates: Start 2020-11-06 (Actual); Primary Completion 2021-09 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
Acceptability of intervention: data directly from web app and survey questions. | Measured at post-intervention (10 weeks)
  Measured through website utilization (e.g. number of visits to app, visit duration, number of steps completed, time spent on each step, number of visits to Routines, time spent at each Routine, Routines marked as favourites by users, ratings of usefulness and challenge of each step) and specific questions (developed by researchers).
Acceptability of intervention: data directly from web app and survey questions. | Measured at post-intervention (6 months)
  Measured through website utilization (e.g. number of visits to app, visit duration, number of steps completed, time spent on each step, number of visits to Routines, time spent at each Routine, Routines marked as favourites by users, ratings of usefulness and challenge of each step) and specific questions (developed by researchers).
Acceptability of study procedures. | Measured at post-intervention (10 weeks)
  Measured through specific questions (developed by researchers) to assess acceptability and proportion of completed online surveys.
  Reasons for non-participation or withdrawal.
Combined demand of intervention and study procedures. | Measured at post-intervention (10 weeks)
  Measured with recruitment and attrition rates (including reported reasons for non-participation or withdrawal).
Combined demand of intervention and study procedures. | Measured at post-intervention (6 months)
  Measured with recruitment and attrition rates (including reported reasons for non-participation or withdrawal).
Implementation of intervention and study procedures reports. | Measured at post-intervention (10 weeks)
  Measured with number of reports of inability to access MyJourney or complete steps or any other questions affecting implementation or reports of problems receiving invitations and accessing the online questionnaires.
Implementation of intervention and study procedures reports. | Measured at post-intervention (6 months)
  Measured with number of reports of inability to access MyJourney or complete steps or any other questions affecting implementation or reports of problems receiving invitations and accessing the online questionnaires.
Practicalities of intervention. | Measured at post-intervention (10 weeks)
  Measured with time for participants to work through all steps in intervention.
Practicalities of intervention. | Measured at post-intervention (6 months)
  Measured with time for participants to work through all steps in intervention.
Practicalities of study procedures. | Measured at post-intervention (10 weeks)
  Measured with length of time for researchers to administer (including time taken to send all required reminders and time taken to respond to emails and respond to queries from participants.
Practicalities of study procedures. | Measured at post-intervention (6 months)
  Measured with length of time for researchers to administer (including time taken to send all required reminders and time taken to respond to emails and respond to queries from participants.
Adaption of study procedures. | Measured at post-intervention (10 weeks)
  Measured with reports of different strategies (e.g. dissemination, recruitment, query resolution) required for Portugal (PT) and United Kingdom (UK).
Adaption of study procedures. | Measured at post-intervention (6 months)
  Measured with reports of different strategies (e.g. dissemination, recruitment, query resolution) required for Portugal (PT) and United Kingdom (UK).
Limited Efficacy Testing - changes from baseline in mental health | From baseline to 10 weeks.
  Measured with the Mental Health Inventory-5 (MHI-5; Veit and Ware, 1983). The total scores range from 1 to 100, with higher scores indicating higher mental health.
Limited Efficacy Testing - changes from baseline in mental health | From baseline to 6 months.
  Measured with the Mental Health Inventory-5 (MHI-5; Veit and Ware, 1983). The total scores range from 1 to 100, with higher scores indicating higher mental health.
Limited Efficacy Testing - changes from baseline in hedonic wellbeing | From baseline to 10 weeks.
  Measured with the World Health Organisation - Five Wellbeing Index (WHO-5; Topp et al., 2015). The total score ranges between 0 to 25, is multiplied by 4 to give the final score, with 0 representing the worst imaginable well-being and 100 representing the best imaginable well-being.
Limited Efficacy Testing - changes from baseline in hedonic wellbeing | From baseline to 6 months.
  Measured with the World Health Organisation - Five Wellbeing Index (WHO-5; Topp et al., 2015). The total score ranges between 0 to 25, is multiplied by 4 to give the final score, with 0 representing the worst imaginable well-being and 100 representing the best imaginable well-being.
Limited Efficacy Testing - changes from baseline in eudaimonic wellbeing | From baseline to 10 weeks.
  Measured with the Office of National Statistics eudaimonic subjective well-being scale (Office of National Statistics, 2012). The total scores range between 0 and 10 with higher scores indicating higher eudaimonic wellbeing.
Limited Efficacy Testing - changes from baseline in eudaimonic wellbeing | From baseline to 6 months.
  Measured with the Office of National Statistics eudaimonic subjective well-being scale (Office of National Statistics, 2012). The total scores range between 0 and 10 with higher scores indicating higher eudaimonic wellbeing.
Limited Efficacy Testing - changes from baseline in posttraumatic growth | From baseline to 10 weeks.
  Measured with the Posttraumatic growth inventory short form (PTG-SF; Cann et al., 2009). The total scores range from 0 to 50, with higher scores indicating higher posttraumatic growth.
Limited Efficacy Testing - changes from baseline in posttraumatic growth | From baseline to 6 months.
  Measured with the Posttraumatic growth inventory short form (PTG-SF; Cann et al., 2009). The total scores range from 0 to 50, with higher scores indicating higher posttraumatic growth.
Limited Efficacy Testing - changes from baseline in happiness | From baseline to 10 weeks.
  Measured with the single item happiness scale (Ahrendt et al., 2017). The total scores range from 1 to 10, with higher scores indicating higher levels of happiness.
Limited Efficacy Testing - changes from baseline in happiness | From baseline to 6 months.
  Measured with the single item happiness scale (Ahrendt et al., 2017). The total scores range from 1 to 10, with higher scores indicating higher levels of happiness.
Limited Efficacy Testing - changes from baseline in satisfaction with life | From baseline to 10 weeks.
  Measured with the single item satisfaction with life scale (Ahrendt et al., 2017). The total scores range from 1 to 10, with higher scores indicating higher satisfaction with life.
Limited Efficacy Testing - changes from baseline in satisfaction with life | From baseline to 6 months.
  Measured with the single item satisfaction with life scale (Ahrendt et al., 2017). The total scores range from 1 to 10, with higher scores indicating higher satisfaction with life.

SECONDARY OUTCOMES:
Changes from baseline in acceptance | From baseline to 10 weeks.
  Measured with the SCREENIVF Questionnaire (partial) (Verhaak et al., 2010). The total score ranges between 6 to 24, with higher scores indicating higher acceptance.
Changes from baseline in self-compassion | From baseline to 10 weeks.
  Measured with the self-compassion scale short form (SCS-SF; Raes et al., 2011). The total score ranges between 1 and 48, with higher scores indicating higher self-compassion.
  Openness to experience subscale-Comprehensive Assessment of Acceptance and Commitment Therapy processes (CompACT) (Francis et al., 2016)
Changes from baseline in openness to experience (acceptance and defusion) | From baseline to 10 weeks.
  Measured with the Openness to experience subscale-Comprehensive Assessment of Acceptance and Commitment Therapy processes (CompACT; Francis et al., 2016). The total score ranges from 0 to 70, with higher scores indicating higher openness to experience.
Changes from baseline in positive reframing coping | From baseline to 10 weeks.
  Measured with the Brief COPE Inventory (partial) (Carver, Scheier, & Weintraub, 1989).The total score ranges from 1 to 16, with higher scores indicating higher positive reframing coping.
  Motivation and activation subscale-CompACT (Francis et al., 2016)
Changes from baseline in valued action | From baseline to 10 weeks.
  Measured with the Motivation and activation subscale-Comprehensive Assessment of Acceptance and Commitment Therapy processes (CompACT; Francis et al., 2016). The total score ranges from 0 to 48, with higher scores indicating higher valued action.
Changes from baseline in goal re-engagement | From baseline to 10 weeks.
  Measured with the goal re-engagement scale (Wrosch, Scheier, Carver, & Schulz, 2003). The total score ranges from 6 and 30, with higher scores indicating greater engagement in other meaningful life goals
  Committed action scale (CAQ-8) (McCracken, Chilcot, & Norton, 2015)
Changes from baseline in committed action | From baseline to 10 weeks.
  Measured with the Committed action scale (CAQ-8; McCracken, Chilcot, & Norton, 2015). The total score ranges from 0 to 48, with higher scores indicating higher committed action.
Changes from baseline in social connection | From baseline to 10 weeks.
  Measured with the Fertility Problem Inventory - social concern subscale (Newton, Sherrard, & Glavac, 1999). The total score ranges from 1 to 60, with higher scores indicating higher perceived social connection.

CONTACTS AND LOCATIONS:
Overall Officials: Beth Rowbottom, Principal Investigator — School of Psychology, Cardiff University; Sofia Gameiro, Principal Investigator — School of Psychology, Cardiff University
Locations (1):
- Cardiff University, Cardiff, United Kingdom

REFERENCES:
- [Background] Gameiro S, Finnigan A. Long-term adjustment to unmet parenthood goals following ART: a systematic review and meta-analysis. Hum Reprod Update. 2017 May 1;23(3):322-337. doi: 10.1093/humupd/dmx001. PMID 28164236
- [Background] Verhaak CM, Lintsen AM, Evers AW, Braat DD. Who is at risk of emotional problems and how do you know? Screening of women going for IVF treatment. Hum Reprod. 2010 May;25(5):1234-40. doi: 10.1093/humrep/deq054. Epub 2010 Mar 13. PMID 20228392
- [Background] Raes F, Pommier E, Neff KD, Van Gucht D. Construction and factorial validation of a short form of the Self-Compassion Scale. Clin Psychol Psychother. 2011 May-Jun;18(3):250-5. doi: 10.1002/cpp.702. Epub 2010 Jun 8. PMID 21584907
- [Background] Francis, A. W., Dawson, D. L., & Golijani-Moghaddam, N. The development and validation of the Comprehensive assessment of Acceptance and Commitment Therapy processes (CompACT). Journal of contextual behavioral science. 2016; 5(3): 134-145.
- [Background] Wrosch C, Scheier MF, Miller GE, Schulz R, Carver CS. Adaptive self-regulation of unattainable goals: goal disengagement, goal reengagement, and subjective well-being. Pers Soc Psychol Bull. 2003 Dec;29(12):1494-508. doi: 10.1177/0146167203256921. PMID 15018681
- [Background] McCracken LM, Chilcot J, Norton S. Further development in the assessment of psychological flexibility: a shortened Committed Action Questionnaire (CAQ-8). Eur J Pain. 2015 May;19(5):677-85. doi: 10.1002/ejp.589. Epub 2014 Sep 2. PMID 25181605
- [Background] Newton CR, Sherrard W, Glavac I. The Fertility Problem Inventory: measuring perceived infertility-related stress. Fertil Steril. 1999 Jul;72(1):54-62. doi: 10.1016/s0015-0282(99)00164-8. PMID 10428148
- [Derived] Rowbottom B, Galhardo A, Donovan E, Gameiro S. Feasibility randomized controlled trial of a self-guided online intervention to promote psychosocial adjustment to unmet parenthood goals. Hum Reprod. 2022 Sep 30;37(10):2412-2425. doi: 10.1093/humrep/deac168. PMID 36001052
- See also: MyJourney website — http://myjourney.pt